CLINICAL TRIAL: NCT05225558
Title: A Multicenter, Double-blinded, Randomized, Parallel Design, Phase IIa Clinical Trial to Evaluate the Efficacy, Safety and PK of LCB01-0371 With Vancomycin Versus Vancomycin Monotherapy in Patients With MRSA Bacteremia
Brief Title: A Phase 2a Study, Effect of Vancomycin With vs Without Delpazolid (LCB01-0371) in Patients With MRSA Bacteremia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination; Difficulties in enrolling subjects due to the decrease in patients with MRSA bacteremia
Sponsor: LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCB35-0371-21-2-01
Record Dates: First submitted 2022-01-26; First posted 2022-02-04 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-03

CONDITIONS: MRSA Bacteremia
Keywords: MRSA; Staphylococcus aureus bacteremia; SAB; bloodstream infection; BSI; Bacteremia
MeSH Terms: conditions — Sepsis; Bacteremia | interventions — delpazolid; Vancomycin

STUDY DESIGN:
Intervention Model Description: Placebo-controlled
Who Masked: Participant, Investigator
Masking Description: Double-blind with placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination therapy - Vancomycin (IV) plus Delpazolid (PO) (Experimental): Vancomycin: IV infusion per 2020 IDSA guideline
  * Intravenous Vancomycin dosed as per 2020 IDSA guideline
  * Doses of 15 to 20 mg/kg (based on actual body weight) administered every 8 to 12 hours as an intermittent infusion were recommended for most patients with normal renal function when assuming a MICBMD of 1 mg/L.
  * Depending on the investigator's judgment, it was allowed to change to Daptomycin after at least one week of administration of Vancomycin, and also it was allowed to change to oral antibiotics other than oxazolidinones after two weeks of administration of Vancomycin (including Daptomycin).
  Delpazolid: 800 mg, BID, PO
  Interventions: Drug: Delpazolid; Drug: Vancomycin
- Monotherapy - Vancomycin (IV) plus Placebo of Delpazolid (PO) (Placebo Comparator): Vancomycin: IV infusion per 2020 IDSA guideline
  * Intravenous Vancomycin dosed as per 2020 IDSA guideline
  * Doses of 15 to 20 mg/kg (based on actual body weight) administered every 8 to 12 hours as an intermittent infusion were recommended for most patients with normal renal function when assuming a MICBMD of 1 mg/L.
  * Depending on the investigator's judgment, it was allowed to change to Daptomycin after at least one week of administration of Vancomycin, and also it was allowed to change to oral antibiotics other than oxazolidinones after two weeks of administration of Vancomycin (including Daptomycin).
  Placebo of Delpazolid: BID, PO
  Interventions: Drug: Vancomycin; Drug: Placebo of Delpazolid

INTERVENTIONS:
Drug: Delpazolid — BID, PO
  Other Names: LCB01-0371
  Arms: Combination therapy - Vancomycin (IV) plus Delpazolid (PO)
Drug: Vancomycin — IV infusion per 2020 IDSA guideline
Drug: Placebo of Delpazolid — BID, PO
  Other Names: Placebo of LCB01-0371
  Arms: Monotherapy - Vancomycin (IV) plus Placebo of Delpazolid (PO)

SUMMARY:
The objectives of this study is to exploratory whether Vancomycin + Delpazolid is more effective to the standard of treatment (Vancomycin)/ for hospitalized adults with MRSA bacteraemia.

DETAILED DESCRIPTION:
The mortality from S aureus bacteremia is higher for MRSA than for methicillin-susceptible S aureus (MSSA), typically at 20% to 25%.

The current standard therapy for MRSA bacteremia is Vancomycin. Vancomycin has many shortcomings, including poor tissue penetration and slow killing time. Vancomycin has reduced efficacy against MRSA and tended to increase the MIC level (called MIC creep). Addition of Delpazolid to Vancomycin could improve the known drawbacks of Vancomycin alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥19 years of age on the date of written consent
* Subject who has confirmed positive MRSA at least one set of blood cultures within 72 hours prior to randomization OR, Subject who has confirmed positive MRSA at least one set of blood culture whthin 96 hours prior to randomization and treated with vancomycin at least 72 hours prior to randomization
* Subject who has clinical symptoms or signs of MRSA bacteremia according to the judgment of the investigator
* Subject who voluntarily decides to participate in this clinical trial after being explained fully, and agrees in writing to implement the clinical trial compliance matters

Exclusion Criteria:

* Subject with polymicrobial bacteremia or infections including Gram-negative strain
* Subject undergoing or in need of treatment with antiviral or antifungal drugs
* Subject who has received treatment for MRSA bacteremia within 3 months of screening (Subjects who have "re-infection" by investigator's judgement may participant in the study.)
* Subject who has been administered effective antibiotics against MRSA (Vancomycin, etc.) for more than 96 hours prior to the first investigational product administration. (However, antibiotics effective for MRSA such as vancomycin are allowed to be administered for less than 72 hours.)
* Septic shock patients
* Subject who has hypersensitivity to vancomycin or linezolid
* Subject who has a history of hypersensitivity to peptide-based antibiotics and aminoglycoside-based antibiotics
* Subject who is receiving a MAO inhibitor(MAOI) or has received MAOI within 14 days of the first investigational drug administration
* Subject taking serotonin reuptake inhibitors, tricyclic antidepressants, serotonin 5-HT1 receptor agonists (triptan), meperidine, or buspirone
* Subject with severely decreased immunity (Severe neutropenia (ANC <0.5×10^9/L) etc.)
* Subject who is expected to die within 2 days due to serious complications of MRSA bacteremia based on the judgment of the investigator
* Body Mass Index (BMI) ≥35 kg/m2
* Subject who is unable to administer drugs orally
* Pregnant or lactating female, female or male with childbearing potential who disagrees with the use of appropriate contraceptive methods during the study and up to 14 days after the last dose of the investigator product
* Subject who has received other clinical trial drugs within 30 days of screening
* Subject who is not suitable for participation in this clinical trial according to the medical findings of investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongbin Kim, Principal Investigator — Seoul National University Bundang Hospital
Locations (6):
- South Korea (6):
  - Chosun University Hospital, Gwangju
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual patient data, that underlie the results in published article(s) based on data from the trial which including text, tables, figures will be presented to various stakeholders. This reported will be presented to various stakeholder during various forums or meetings. First results will be disclosed to participants, staff and our site Community Advisory Board. Thereafter we would invite several stakeholders from the community or visit their establishments to review study results. Simultaneously, the studying findings report will be sent to the various regulatory authorities, including the National Department of Health (NDoH). With NDoH and its divisions we will establish needs for further engagement and suggestions for policy or programmatic changes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be provided 1-2 years after and up to 5 years after the publication of the article on the results of the trial.
Access Criteria: IPD access will be provided for analyses of the related to the aims of research described in the protocol and for individual patient data meta analyses to researches who provide a methodologically sound proposal to lcb_pv@legochembio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was initiated on 26 Apr 2022 (first signed informed consent) with the date of last participant who completed last study visit on 18 Mar 2024.
  A total of 45 participants were screened. Of these, 40 participants were randomized to 1 of 2 arms. The remaining 5 participants were considered to have been screen failures.
Groups:
- Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID: Vancomycin: IV infusion per 2020 IDSA guideline
  * Intravenous Vancomycin dosed as per 2020 IDSA guideline
  * Doses of 15 to 20 mg/kg (based on actual body weight) administered every 8 to 12 hours as an intermittent infusion were recommended for most patients with normal renal function when assuming a MICBMD of 1 mg/L.
  * Depending on the investigator's judgment, it was allowed to change to Daptomycin after at least one week of administration of Vancomycin, and also it was allowed to change to oral antibiotics other than oxazolidinones after two weeks of administration of Vancomycin (including Daptomycin).
  Delpazolid: BID, PO
- Monotherapy - Vancomycin IV Plus Placebo of Delpazolid: Vancomycin: IV infusion per 2020 IDSA guideline
  * Intravenous Vancomycin dosed as per 2020 IDSA guideline
  * Doses of 15 to 20 mg/kg (based on actual body weight) administered every 8 to 12 hours as an intermittent infusion were recommended for most patients with normal renal function when assuming a MICBMD of 1 mg/L.
  * Depending on the investigator's judgment, it was allowed to change to Daptomycin after at least one week of administration of Vancomycin, and also it was allowed to change to oral antibiotics other than oxazolidinones after two weeks of administration of Vancomycin (including Daptomycin).
  Placebo of Delpazolid: BID, PO
Period: Overall Study
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Started | 20 | 20
Safety Set (The safety set consists of all subjects who have received at least one dose of the investigational product.) | 18 | 20
Completed | 10 | 13
Not Completed | 10 | 7
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Adverse Event | 1 | 0
Not completed — If the following treatment failure criteria are met during treatment period | 1 | 2
Not completed — When investigators decide that the subject should stop participating in the trial for other reasons | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety Set (SS)
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 15
  >=65 years | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (9.68) | 64.5 (16.47) | 66.8 (13.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 11 | 10 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Childbearing potential [Count of Participants; unit: Participants] — Population: Only female
  Participants
    number analyzed (Participants) | 7 | 10 | 17
    Yes | 0 | 2 | 2
    No | 7 | 8 | 15
Height (cm) [Mean (Standard Deviation); unit: cm] | 164.15 (6.302) | 161.85 (7.582) | 162.94 (7.009)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 64.77 (9.536) | 63.59 (13.256) | 64.14 (11.506)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 24.020 (3.1754) | 24.229 (4.6732) | 24.130 (3.9823)
Primary Lesion [Count of Participants; unit: Participants] — Multiple counts are possible.
  Participants
    Skin and soft tissue infection | 1 | 6 | 7
    Primary blood stream infection | 1 | 3 | 4
    Native osteoarticular | 2 | 1 | 3
    Intravenous line related | 2 | 7 | 9
    Pleuropulmonary infection | 3 | 0 | 3
    Device related | 0 | 1 | 1
    Infective endocarditis | 2 | 0 | 2
    Unknown | 2 | 0 | 2
    Other | 5 | 3 | 8
Primary lesion removable [Count of Participants; unit: Participants]
  Yes | 7 | 11 | 18
  No | 11 | 9 | 20
Primary lesion removed [Count of Participants; unit: Participants] — Population: If the primary lesion removable is 'Yes'
  Participants
    number analyzed (Participants) | 7 | 11 | 18
    Yes | 4 | 6 | 10
    No | 3 | 5 | 8
Vancomycin MIC [Count of Participants; unit: Participants] — Evaluation of the MIC (Minimum Inhibitory Concentration) of vancomycin was performed the time of screening when deemed necessary by the investigator, based on the MIC assessment method established at the site to confirm susceptibility, determine resistance to MRSA, and adjust the vancomycin dose.
  Participants
    <1.5 mcg/mL | 10 | 13 | 23
    ≥1.5 mcg/mL | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Cure Rate at Day 14 After the Start of Treatment (Composite Response Rate: Clinical Improvement Plus Clearance of Bacteremia)_FAS
Description: * 'Overall cure' means that there are no symptoms of infection that existed when enrolled in the clinical trial, there are no new metastatic infection due to MRSA and no new infection (clinical improvement), and MRSA negative is confirmed twice in a row as a result of blood culture tests (clearance of bacteremia). If negative in the blood culture test is confirmed for the first time, additional test will be performed the next day, and if it results negative for a total of two times in a row, it is judged as 'clearance of bacteremia'.
  * Composite Response rate = (number of participants showing overall cure at Day 14/number of participants in each treatment group) x 100
Time Frame: at Day 14
Population: FAS (Full analysis set) : The analysis was conducted on patients who received the IP at least once after randomization and had at least one valid efficacy evaluation result. Additionally, participants who violated the inclusion/exclusion criteria were excluded from the FAS analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 15 | 19
Participants | 9 | 10

2. Primary Outcome: Overall Cure Rate at Day 14 After the Start of Treatment (Composite Response Rate: Clinical Improvement Plus Clearance of Bacteremia)_PPS
Description: as for outcome 1
Time Frame: at Day 14
Population: PPS(Per protocol set): The analysis was conducted on patients from the FAS who completed the study without experiencing major Protocol deviation and whose IP treatment compliance* was less than 80% up to 14 days after the first dose of the IP. Participants whose reason for withdrawal is "Treatment failure criteria are met during the treatment period" are not excluded from the PPS.
  *(Sum of the number (tab) of actually taken up to the 14th day /14 days (minimum administration period)X4(tab))X100
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 11 | 14
Participants | 9 | 9

3. Secondary Outcome: Overall Cure Rate by End of Treatment (EOT)_FAS
Description: as for outcome 1
Time Frame: Day 7 visit and EOT (up to 6 weeks) visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 15 | 19
Participants
  Day 7 | 7 | 6
  End of Treatment | 12 | 14

4. Secondary Outcome: Overall Cure Rate by End of Treatment (EOT)_PPS
Description: as for outcome 1
Time Frame: Day 7 visit and EOT (up to 6 weeks) visit
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 11 | 14
Participants
  Day 7 | 6 | 5
  End of Treatment | 10 | 12

5. Secondary Outcome: Mortality From MRSA Bacteremia by EOT_FAS
Description: * Proportion of participants who died due to MRSA bacteremia
  * Overall mortality = (number of participants who died/number of participants in each treatment group) x 100
Time Frame: During the treatment period (from the first administration to EOT (up to 6 weeks))
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 15 | 19
Participants
  Overall death | 0 | 1
  Death from MRSA bacteremia | 0 | 0

6. Secondary Outcome: Mortality From MRSA Bacteremia by EOT_PPS
Description: as for outcome 5
Time Frame: During the treatment period (from the first administration to EOT (up to 6 weeks))
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 11 | 14
Participants
  Overall death | 0 | 1
  Death from MRSA bacteremia | 0 | 0

7. Secondary Outcome: Relapse Rate of MRSA bacteremia_FAS
Description: * Defined as a positive blood culture to MRSA when previous ones were negative
  * Relapse rate of MRSA bacteremia = (number of participants with Relapse of MRSA bacteremia after clearance of MRSA bacteremia until TOC visit/number of participants with clearance of MRSA bacteremia in each treatment group) x 100
Time Frame: from the first administration to TOC (4 weeks after EOT)
Population: * Participants in FAS who had MRSA negative two consecutive set in the blood culture test
  * FAS (Full analysis set) : The analysis was conducted on participants who received the IP at least once after randomization and had at least one valid efficacy evaluation result. Additionally, participants who violated the inclusion/exclusion criteria were excluded from the FAS analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 15 | 17
Participants | 2 | 1

8. Secondary Outcome: Relapse Rate of MRSA bacteremia_PPS
Description: as for outcome 7
Time Frame: from the first administration to TOC (4 weeks after EOT)
Population: * Participants in PPS who had MRSA negative two consecutive set in the blood culture test
  * PPS (Per protocol set): The analysis was conducted on patients from the FAS who completed the study without experiencing major Protocol deviation and whose IP treatment compliance was less than 80% up to 14 days after the first dose of the IP. Participants whose reason for withdrawal is "Treatment failure criteria are met during the treatment period" are not excluded from the PPS.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 11 | 13
Participants | 2 | 1

9. Secondary Outcome: Clearance Rate of MRSA Bacteremia at Day 3, Day 5, Day 7, Day 14, EOT_FAS
Description: * Proportion of participants who confirmed MRSA negative two consecutive set in the blood culture test
  * Clearance Rate = (number of subjects who achieved clearance at each visit/number of subjects in each treatment group) x 100
Time Frame: Day 3, Day 5, Day 7, Day 14, EOT (up to 6 weeks)
Population: FAS (Full analysis set) : The analysis was conducted on participants who received the IP at least once after randomization and had at least one valid efficacy evaluation result. Additionally, participants who violated the inclusion/exclusion criteria were excluded from the FAS analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 15 | 19
Participants
  Day3: number analyzed (Participants) | 14 | 18
  Day3 | 8 | 6
  Day5: number analyzed (Participants) | 13 | 18
  Day5 | 9 | 11
  Day7: number analyzed (Participants) | 13 | 17
  Day7 | 7 | 6
  Day14: number analyzed (Participants) | 11 | 14
  Day14 | 9 | 11
  End of Treatment | 12 | 14

10. Secondary Outcome: Clearance Rate of MRSA Bacteremia at Day 3, Day 5, Day 7, Day 14, EOT_PPS
Description: as for outcome 9
Time Frame: Day 3, Day 5, Day 7, Day 14, EOT (up to 6 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 11 | 14
Participants
  Day3: number analyzed (Participants) | 10 | 14
  Day3 | 5 | 5
  Day5 | 8 | 8
  Day7 | 6 | 5
  Day14: number analyzed (Participants) | 11 | 13
  Day14 | 9 | 10
  End of Treatment | 10 | 12

11. Secondary Outcome: Persistent Rate of Bacteremia at Day 3, Day 5, Day 7, Day 14_FAS
Description: * Proportion of participants who have positive results on blood culture tests
  * Persistent rate of bacteremia = (number of subjects who showing persistent bacteremia up to each visit /number of subjects in each treatment group up to each visit) x 100
Time Frame: Day 3, Day 5, Day 7, Day 14
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 15 | 19
Participants
  Day3: number analyzed (Participants) | 14 | 18
  Day3 | 6 | 12
  Day5: number analyzed (Participants) | 13 | 18
  Day5 | 4 | 7
  Day7: number analyzed (Participants) | 13 | 17
  Day7 | 1 | 3
  Day14: number analyzed (Participants) | 11 | 14
  Day14 | 0 | 2

12. Secondary Outcome: Persistent Rate of Bacteremia at Day 3, Day 5, Day 7, Day 14_PPS
Description: as for outcome 11
Time Frame: Day 3, Day 5, Day 7, Day 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 11 | 14
Participants
  Day3: number analyzed (Participants) | 10 | 14
  Day3 | 5 | 9
  Day5 | 3 | 6
  Day7 | 0 | 3
  Day14: number analyzed (Participants) | 11 | 13
  Day14 | 0 | 2

13. Secondary Outcome: Time to Clearance of MRSA bacteremia_FAS
Description: If negative in the blood culture test is confirmed for the first time, additional test will be performed the next day, and if it results negative for a total of two times in a row, it is judged as clearance of bacteremia. The period until the clearance of bacteremia is defined as the period (day) from the date of the first blood culture test within 72 hours prior to randomization with MRSA positive (index blood culture) to the date of the blood culture test with the first negative result confirmed.
Time Frame: by EOT (up to 6 weeks)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 15 | 19
days | 7.00 [3.00 to 14.00] | 8.00 [4.00 to 18.00]

14. Secondary Outcome: Time to Clearance of MRSA bacteremia_PPS
Description: as for outcome 13
Time Frame: by EOT (up to 6 weeks)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 11 | 14
days | 4.00 [3.00 to 14.00] | 7.00 [4.00 to 18.00]

15. Other Pre Specified Outcome: Vancomycin MIC Level
Description: Vancomycin minimum inhibitory concentration (MIC) levels
Time Frame: at Screening visit (baseline)
Population: Participants who received the IP at least once and had samples collected for MIC evaluation among the 40 randomized participants.
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 16 | 16
mcg/ml | 0.78 (0.256) | 0.75 (0.258)

16. Other Pre Specified Outcome: Delpazolid MIC Levels
Description: Delpazolid minimum inhibitory concentration (MIC) level by broth microdilution (BMD)
Time Frame: Screening (Baseline), Day 14, EOT
Population: Participants in the Safety Set who were evaluated for Delpazolid MIC at baseline, Day 14, and EOT.
  Of the subjects in the SS (combination: 18 subjects, monotheray: 20 subjects), Delpazolid MIC was evaluated in 18 and 17 subjects from the combination and monotherapy groups at screening, 1 and 2 at Day 14, and 1 and 0 at EOT, respectively.
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
Number analyzed (Participants) | 18 | 20
mcg/ml
  Baseline: number analyzed (Participants) | 18 | 17
  Baseline | 1.1 (0.34) | 1.1 (0.42)
  Day14: number analyzed (Participants) | 1 | 2
  Day14 | 1.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant | 1.0 (0.00)
  End of Treatment: number analyzed (Participants) | 1 | 0
  End of Treatment | 1.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |

17. Other Pre Specified Outcome: Pharmacokinetics (PK) parameters_AUC,ss
Description: Plasma LCB01-0371 concentration data in MRSA bacteremia patients were used to establish a pharmacokinetic model using NONMEM®. A two-compartment model, in which the Hemodialysis (HD) status and albumin as a covariate, was selected as the final model.
  (AUC,ss: Area under the concentration-time curve at steady state)
Time Frame: Plasma samples for pharmacokinetic evaluation were collected once at each timepoint on Day 1 and between Day 3 and end of treatment (EOT), specifically at 30 minutes to 1 hour and 2 to 8 hours after administration of the investigational product.
Population: Out of the total 40 enrolled patients, the blood concentrations of LCB01-0371 from the 15 patients in the treatment group who received LCB01-0371 (excluding the 19 control subjects who received placebo) were included in the population PK model analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Total: Out of the total 40 enrolled patients, the blood concentrations of LCB01-0371 from the 15 patients in the treatment group who received LCB01-0371 (excluding the 19 control subjects who received placebo) were included in the population PK model analysis.
- No ESRD: Subjects without End-Stage Renal Disease (ESRD) based on their medical history
- ESRD: Subjects with End-Stage Renal Disease (ESRD) based on their medical history
- Not Undergoing HD: Subjects without ESRD or Subject with ESRD not undergoing Hemodialysis (HD) based on their medical history
- Undergoing HD: Subjects with ESRD undergoing Hemodialysis (HD) receiving based on their medical history
- No HI/LC: Subjects not included in either LC* or HI** *LC: Liver cirrhosis
  **HI: Hepatic impairment status according to the NCI-ODWG criteria
- HI/LC: Subjects included in either LC* or HI**, i.e., the combination of LC and HI *HI: Hepatic impairment status according to the NCI-ODWG criteria
  **LC: Liver cirrhosis
Arm/Group | Total | No ESRD | ESRD | Not Undergoing HD | Undergoing HD | No HI/LC | HI/LC
Number analyzed (Participants) | 15 | 8 | 7 | 9 | 6 | 10 | 5
ng*h/mL | 90,855.222 (88,895.538) | 83,671.053 (75,411.511) | 99,065.701 (107,966.645) | 112,462.317 (111,518.903) | 58,444.580 (11,292.560) | 59,842.551 (26,423.362) | 152,880.564 (137,383.144)

18. Other Pre Specified Outcome: Pharmacokinetics (PK) parameters_Cmax,ss
Description: Plasma LCB01-0371 concentration data in MRSA bacteremia patients were used to establish a pharmacokinetic model using NONMEM®. A two-compartment model, in which the Hemodialysis (HD) status and albumin as a covariate, was selected as the final model.
  (Cmax,ss: Maximum concentration of drug at steady state)
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Total | No ESRD | ESRD | Not Undergoing HD | Undergoing HD | No HI/LC | HI/LC
Number analyzed (Participants) | 15 | 8 | 7 | 9 | 6 | 10 | 5
ng/mL | 8,595.050 (7,229.136) | 8,610.266 (5,715.031) | 8,577.661 (9,156.152) | 10,903.652 (8,712.950) | 5,132.147 (938.601) | 6,216.075 (1,624.925) | 13,353.002 (11,598.454)

19. Other Pre Specified Outcome: Pharmacokinetics (PK) parameters_Cmin,ss
Description: Plasma LCB01-0371 concentration data in MRSA bacteremia patients were used to establish a pharmacokinetic model using NONMEM®. A two-compartment model, in which the Hemodialysis (HD) status and albumin as a covariate, was selected as the final model.
  (Cmin,ss: Minimum concentration of drug at steady state)
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Total | No ESRD | ESRD | Not Undergoing HD | Undergoing HD | No HI/LC | HI/LC
Number analyzed (Participants) | 15 | 8 | 7 | 9 | 6 | 10 | 5
ng/mL | 6,586.689 (7,255.844) | 5,541.150 (6,209.527) | 7,781.590 (8,644.985) | 7,955.430 (9,284.244) | 4,533.576 (1,032.638) | 3,992.895 (2,331.779) | 11,774.277 (11,026.039)

20. Other Pre Specified Outcome: Pharmacokinetics (PK) parameters_Tmax,ss
Description: Plasma LCB01-0371 concentration data in MRSA bacteremia patients were used to establish a pharmacokinetic model using NONMEM®. A two-compartment model, in which the Hemodialysis (HD) status and albumin as a covariate, was selected as the final model.
  (Tmax,ss: Time to reach Cmax at steady state)
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Total | No ESRD | ESRD | Not Undergoing HD | Undergoing HD | No HI/LC | HI/LC
Number analyzed (Participants) | 15 | 8 | 7 | 9 | 6 | 10 | 5
h | 3.562 (1.322) | 3.083 (1.515) | 4.110 (0.861) | 3.286 (1.542) | 3.978 (0.861) | 3.291 (1.429) | 4.105 (0.984)

21. Other Pre Specified Outcome: Pharmacokinetics (PK) parameters_t1/2β
Description: Plasma LCB01-0371 concentration data in MRSA bacteremia patients were used to establish a pharmacokinetic model using NONMEM®. A two-compartment model, in which the Hemodialysis (HD) status and albumin as a covariate, was selected as the final model.
  (t1/2β : Terminal elimination half-life)
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Total | No ESRD | ESRD | Not Undergoing HD | Undergoing HD | No HI/LC | HI/LC
Number analyzed (Participants) | 15 | 8 | 7 | 9 | 6 | 10 | 5
h | 9,292.011 (28,745.858) | 1,689.649 (4,369.248) | 17,980.425 (41,721.541) | 13,973.252 (37,076.761) | 2,270.149 (3,949.333) | 425.392 (572.107) | 27,025.249 (47,976.785)

22. Other Pre Specified Outcome: Pharmacokinetics (PK) parameters_MRT,ss
Description: Plasma LCB01-0371 concentration data in MRSA bacteremia patients were used to establish a pharmacokinetic model using NONMEM®. A two-compartment model, in which the Hemodialysis (HD) status and albumin as a covariate, was selected as the final model.
  (MRT,ss: Mean residence time at steady state)
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Total | No ESRD | ESRD | Not Undergoing HD | Undergoing HD | No HI/LC | HI/LC
Number analyzed (Participants) | 15 | 8 | 7 | 9 | 6 | 10 | 5
h | 6,843.719 (20,060.037) | 1,159.389 (3,024.815) | 13,340.095 (28,912.833) | 9,730.567 (25,868.738) | 2,513.446 (4,304.084) | 436.814 (654.947) | 19,657.528 (33,160.057)

ADVERSE EVENTS:
Time Frame: From IP administration to TOC (Test of Cure, 4 weeks after EOT*), approximately 10 weeks *EOT (End of treatment): up to 6 weeks
Description: All clinically significant medical conditions or abnormalities observed from the administration of the IP until TOC were collected as AEs.
  If an AE identified before the administration of the IP worsened in severity after the IP administration, it was collected as a new AE.
Arm/Group | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/20
Other Adverse Events (participants affected / at risk) | 13/18 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID (N=18) | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid (N=20)
end stage renal disease (Renal and urinary disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy - Vancomycin IV Plus Delpazolid 800 mg, PO, BID (N=18) | Monotherapy - Vancomycin IV Plus Placebo of Delpazolid (N=20)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Melaena 0 [0] 2 (10.00) [2] (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (7)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Escherichia test positive (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (4) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial rupture (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT05225558/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT05225558/SAP_001.pdf